CLINICAL TRIAL: NCT04066062
Title: Registry of Coronary Computed Tomography Angiography Intravenous Ultrasound and Optical Coherence Tomography to Compare Invasive/Non-invasive Imaging Modalities for Determination of Severity Volume and Type of Coronary Atherosclerosis
Brief Title: Multicentre Registry of CCTA, IVUS and OCT
Status: Active, not recruiting | Type: Observational
Sponsor: Cleerly, Inc. (Industry)
Collaborators: Toho University - Omori Medical Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: Invictus Registry
Record Dates: First submitted 2019-08-15; First posted 2019-08-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease
Keywords: CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: A total of 700 vessel from 700 patients clinically indicated CCTA and IVUS or OCT performed within 3 months.
- Prospective: A total of 1,000 subjects will be enrolled in this Registry. This number of subject is expected to provide a maximum of 1,300 vessels. All CCTA and IVUS/OCT will be performed within 3 months

SUMMARY:
The Invictus Registry will compare the diagnostic performance of coronary computed tomography angiography (CCTA) versus intravascular imaging by intravenous ultrasound (IVUS) or optical coherence tomography (OCT) for the measurement of minimum lumen area, the identification of stenosis severity, burden, morphology and vulnerability of coronary atherosclerosis.

DETAILED DESCRIPTION:
Clinical Significance:

Coronary computed tomographic angiography (CCTA) is a robust non-invasive modality to evaluate the presence, extent and severity of Coronary Artery Disease (CAD). For a plaque assessment, previous studies demonstrated that CCTA provides a high correlation with intravascular imaging by intravenous ultrasound (IVUS) in assessing coronary plaque characteristics stenosis severity and volume. High risk (vulnerable) plaque characteristics (positive remodeling, low attenuation plaque, spotty calcifications) are recognized to be more prone to rupture with increased rates of short-term cardiovascular disease events. Although several studies similarly demonstrated the good concordance between CCTA and IVUS or optical coherence tomography (OCT) in assessing high risk plaque features, patient numbers in these prior studies were limited to fully understand the effect of CCTA for the assessment of coronary atherosclerotic plaque features.

The Research is a multi-center, registry enrolling patients with single/multi vessel atherosclerotic coronary artery disease. The study will be conducted in up to 15 Medical Centers in Japan. In each patient, a CCTA, IVUS), and/ or OCT will be performed, to provide a total of 1,300 vessels from 1,000 patients. Thus, the full cohort (Prospective plus Retrospective patients) will provide a total of 2,000 vessels as basis for a diagnostic performance comparison between CCTA and IVUS or OCT. Accrual is expected to take 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, inclusive of release of medical information, and Health Insurance Portability and Accountability Act (HIPAA) documentation
* Age 18 years or older
* Known or suspected Coronary Artery Disease and subsequently indicated for coronary artery angiography

Exclusion Criteria:

* Individuals unable to provide informed consent
* Acute ST elevation myocardial infarction
* Pregnant woman
* Angiographically visible thrombus at the site of the lesion interrogated by IVUS or OCT
* Patients with lesions required balloon angioplasty before OCT and/or IVUS

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with single/multi vessel atherosclerotic coronary artery disease
Sampling Method: Probability Sample
Enrollment: 1700 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare the diagnostic performance of CCTA versus IVUS or OCT for the measurement of minimum lumen area. | June 2019- June 2021
  Patients will undergo invasive coronary angiography with IVUS/OCT for the measurement of minimum lumen area, the identification of stenosis severity, burden, morphology and vulnerability of coronary atherosclerosis.
  The co-registration of IVUS/OCT images with CCTA segmented images will be implemented in the following three stages by locating the corresponding anatomical landmarks/fiduciary points (coronary ostia, side-branches, calcified plaques, and/or overlapping veins) and matching the corresponding coronary segments in all the imaging modalities

CONTACTS AND LOCATIONS:
Overall Officials: Rine Nakanishi, MD, Principal Investigator — Toho University - Omori Medical Center
Locations (9):
- Japan (9):
  - Ehime University, Ehime
  - Hiroshima University, Hiroshima
  - Yotsuba Circulation Clinic, Matsuyama
  - Okayama Red Cross Hospital, Okayama
  - Toho University Omori Medical Center, Tokyo
  - Edogawa Hospital, Tokyo
  - Juntendo University, Tokyo
  - Sakakibara Heart Institute, Tokyo
  - Tokai University, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nakanishi R, Okubo R, Sobue Y, Kaneko U, Sato H, Fujimoto S, Nozaki Y, Kajiya T, Miyoshi T, Ichikawa K, Abe M, Kitagawa T, Ikenaga H, Osawa K, Saji M, Iguchi N, Nakazawa G, Takahashi K, Ijich T, Mikamo H, Kurata A, Moroi M, Iijima R, Malkasian S, Crabtree T, Chamie D, Alexandra LJ, Min JK, Earls JP, Matsuo H. Rationale and design of the INVICTUS Registry: (Multicenter Registry of Invasive and Non-Invasive imaging modalities to compare Coronary Computed Tomography Angiography, Intravascular Ultrasound and Optical Coherence Tomography for the determination of Severity, Volume and Type of coronary atherosclerosiS). J Cardiovasc Comput Tomogr. 2023 Nov-Dec;17(6):401-406. doi: 10.1016/j.jcct.2023.08.011. Epub 2023 Sep 9. PMID 37679247